CLINICAL TRIAL: NCT04517097
Title: Study of the Specific Seroprevalence of SARS-CoV-2 in a Sample of Patients and Salaried Staff From a French Anti-cancer Center at the End of the Containment Period of the SARS-CoV-2 Pandemic
Acronym: canSEROcov
Status: Completed | Type: Observational
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-A00877-32
Record Dates: First submitted 2020-08-14; First posted 2020-08-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Cancer
Keywords: SARS-CoV-2; seroprevalence
MeSH Terms: conditions — Neoplasms | interventions — Blood Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patient group: patients treated in the french anti-cancer center of the study
  Interventions: Biological: blood sample
- salaried staff group: all salaried staff of the french anti-cancer center of the study
  Interventions: Biological: blood sample

INTERVENTIONS:
Biological: blood sample — one blood sample and one questionnaire to each patient and salaried staff included
  Other Names: questionnaire

SUMMARY:
Since March 2020, France has been confronted with the SARS-COV-2 pandemic. Analysis of the data of its spread would indicate that close contact between individuals is necessary and containment would be the best way to contain this virus. France has therefore been contained since March 17, 2020 until 11 May 2020.

In order to assess the impact of the measures taken (containment) to protect patients and salaried staff of a french anti-cancer center on the spread of the virus, this observational study assesses the specific seroprevalence of SARS-COV-2 in all caregivers and non-carers of this hospital and in patients treated in consultation, day hospitalization, full hospitalization at the end of the containment period.

The objective for the staff cohort is to describe the seroprevalence and the link between the seroprevalence and sociological / demographic factors relating to the category of profession, to the contacts with the patients, to the presence in the hospital during the period of containment, to the conditions of home containment.

The objective for the patient cohort is to describe the seroprevalence and the link between the seroprevalence and factors relating to the type of cancer treated, the type of treatment and their possible modification during the period of containment, to the conditions of home containment.

ELIGIBILITY:
Inclusion Criteria:

* Patient group:

Patient over 18 years old. Patient who gave his non-opposition to carrying out the study. Patient affiliated to the social security scheme.

* Salaried staff group:

Salaried staff over 18 years old. Salaried staff not opposing the carrying out of the study. Salaried staff affiliated to the social security scheme.

Exclusion Criteria:

* Patient group:

Minor patient, under legal protection or subject to a legal protection measure Patient deprived of liberty or under guardianship Inability to undergo medical monitoring of the trial for geographical, social or psychological reasons Patient refusal to participate Pregnant or nursing mothers

* Salaried staff group:

Underage salaried staff or under legal protection Salaried staff deprived of liberty or under guardianship Inability of the salaried staff to submit to the monitoring of the test: filling out the questionnaire and taking a blood sample Salaried staff refusal to participate in the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients treated in the anti-cancer hospital of the study and all salaried staff of the anti-cancer hospital of the study.
Sampling Method: Probability Sample
Enrollment: 1680 (Actual)
Dates: Start 2020-05-12 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
seroprevalence of SARS-CoV-2 | inclusion
  rate of specific SARC-Cov-2 IgM and IgG

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Georges-François LECLERC, Dijon, France

IPD SHARING:
Plan to Share IPD: Undecided